CLINICAL TRIAL: NCT07201389
Title: A Study to Investigate DigniCap Scalp Cooling on Black Patients for Prevention of Chemotherapy-induced Alopecia.
Brief Title: CARE (Chemotherapy Alopecia REduction)
Acronym: CARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Pavani Chalasani, Professor of Medicine; Director, Division of Hematology Oncology, George Washington University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARE (Scalp Cooling Protocol)
Record Dates: First submitted 2025-09-24; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Breast - Female; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III; Chemotherapy Induced Alopecia
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Scalp Cooling Arm (Experimental): DigniCap Scalp Cooling will be applied to all participants undergoing chemotherapy
  Interventions: Device: Scalp Cooling by DigniCap

INTERVENTIONS:
Device: Scalp Cooling by DigniCap — Scalp cooling with the DigniCap Delta will occur with each chemotherapy dose. The cooling wrap is primed, fitted, and checked for proper contact before a standardized pre-cool phase of 20-30 minutes. Cooling continues during chemotherapy, followed by a post-cool phase of 90-180 minutes based on regimen. The system circulates temperature-controlled coolant through channels in the wrap, with sensors monitoring flow and scalp temperature; a safety sensor ensures scalp temperature never falls below 32°F (0°C). Alerts notify staff of low flow or temperature issues. After cooling, the cap is loosened for 5 minutes to warm before removal, and subjects are given 5 minutes to acclimate before standing.

SUMMARY:
The goal of this research study is to determine if the DigniCap Scalp Cooling System can help prevent chemotherapy-induced hair loss in Black patients.

DETAILED DESCRIPTION:
The purpose of this study is to assess whether the DigniCap Scalp Cooling System can help prevent chemotherapy-induced hair loss in Black patients undergoing treatment for breast cancer. The primary objective of this study is to provide a preliminary assessment of the efficacy of the DigniCap Scalp Cooling in Black patients as prevention for chemotherapy induced alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with early stage breast cancer (stage I-III)
* Self-identify as Black
* Planned therapy with taxane and/or anthracycline-based chemotherapy (at least 4 cycles must be planned)

  -≥ 21 years of age
* Able to give informed consent

Exclusion Criteria:

* Female pattern hair loss or hair loss disorder
* Scalp folliculitis
* Scalp psoriasis Scalp seborrheic dermatitis
* Inflammatory scalp conditions such as lichen planopillaris or alopecia areata
* Subjects wearing wigs or subjects who shave their hair prior to chemotherapy
* Unable to provide consent or make allotted clinical visits
* Subjects with cold agglutinin disease or cold urticaria
* Unwilling to remove hair extensions during treatment phase which can interfere with study assessments
* History or whole brain irradiation
* History of prior systemic chemotherapy

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Black women, black female
Enrollment: 30 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Success in hair preservation after at least four cycles of chemotherapy | From enrollment to the end of study (2 years)
  Success is defined as CTCAE v5.0 alopecia grade 0 (no hair loss) or grade 1 (<50% hair loss not requiring a wig). Failure is defined as CTCAE v5.0 grade 2 (≥50% hair loss, requiring use of a wig) or higher.

SECONDARY OUTCOMES:
To estimate participant reported comfort of using Digniticap | From enrollment to the end of study (2 years)
  Participants will be asked if they find the procedure acceptable or unacceptable based on comfort scale used in Massey study (2004). The scale range:
  Question for participant: How comfortable were you in general throughout the scalp cooling period?
  Scale:
  1. Very Comfortable
  2. Reasonably Comfortable
  3. Comfortable
  4. Uncomfortable
  5. Very Uncomfortable
Evaluate quality of life (QOL) during study treatment phase- HADS | From enrollment to the end of study (2 years)
  QOL will be assessed by the HADS (anxiety summary and depression summary). It will be administered at baseline, after 4 cycles (except if someone is on weekly regimen, then the assessments will be done every 2 weeks x 4 times) and then after completion of chemotherapy (if the subject is receiving more than 4 cycles).
  1.The HADS will be used to assess anxiety and depression. It includes 7 questions to assess anxiety and 7 to assess depression. The summary scores (sum of the 7 question items) for anxiety and depression range from 0 to 21: scores of 0 to 7 are considered normal, 8 to 10 are considered borderline abnormal (borderline case), and 11 to 21 are considered abnormal (case).
Evaluate quality of life (QOL) during study treatment phase- BIS | From enrollment to the end of study (2 years)
  QOL will be assessed by the BIS (body image scale appendix included protocol). It will be administered at baseline, after 4 cycles (except if someone is on weekly regimen, then the assessments will be done every 2 weeks x 4 times) and then after completion of chemotherapy (if the subject is receiving more than 4 cycles).
  1. The BIS summary score will be the sum of the first 9 (of 10) items in the BIS. The summary score ranges from 0 to 27; a score of 0 indicates no symptoms or distress, and a higher score indicates increasing symptoms or distress.

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington-Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dilawari A, Gallagher C, Alintah P, Chitalia A, Tiwari S, Paxman R, Adams-Campbell L, Dash C. Does Scalp Cooling Have the Same Efficacy in Black Patients Receiving Chemotherapy for Breast Cancer? Oncologist. 2021 Apr;26(4):292-e548. doi: 10.1002/onco.13690. Epub 2021 Feb 17. PMID 33512741
- [Background] Benjamin B, Ziginskas D, Harman J, Meakin T. Pulsed electrostatic fields (ETG) to reduce hair loss in women undergoing chemotherapy for breast carcinoma: a pilot study. Psychooncology. 2002 May-Jun;11(3):244-8. doi: 10.1002/pon.593. PMID 12112485
- [Background] Pozo-Kaderman C, Kaderman RA, Toonkel R. The psychosocial aspects of breast cancer. Nurse Pract Forum. 1999 Sep;10(3):165-74. PMID 10614362